CLINICAL TRIAL: NCT02162654
Title: The Role of Remote Ischemic Preconditioning in the Prevention of Ischemic Brain Damage During Intracranial Aneurysm Treatment (RIPAT) - A Prospective Randomized Exploratory Study
Brief Title: Remote Ischemic Preconditioning for Intracranial Aneurysm Treatment
Acronym: RIPAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Martin Ortler, MD MSc, Vice Chairman, Clinical Department of Neurosurgery, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20131101-823
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Cerebral Aneurysm
Keywords: neuroprotection; ischemic preconditioning; cerebral aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote ischemic preconditioning (Active Comparator): Inflation of a blood pressure cuff around an arm with the patient under general anesthesia prior to start aneurysm treatment
  Interventions: Procedure: Remote ischemic preconditioning
- Sham preconditioning (Sham Comparator): Sham inflation of a blood pressure cuff around an arm with the patient under general anesthesia prior to start aneurysm treatment
  Interventions: Procedure: Sham preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — The blood pressure cuff is inflated to 200 mmHg for 3 x 5 minutes with 5 minutes of reperfusion by complete cuff deflation each.
  Arms: Remote ischemic preconditioning
Procedure: Sham preconditioning — The blood pressure cuff is inflated to 10 mmHg for 3 x 5 minutes with 5 minutes of complete cuff deflation each.
  Arms: Sham preconditioning

SUMMARY:
The RIPAT study is a prospective, randomized, double-blind study organized by the neurovascular group of the Clinical Department of Neurosurgery of Innsbruck Medical University, Innsbruck, Austria. Patients aged 18+ in whom the treatment of an un-ruptured intracranial aneurysm is indicated are eligible for study participation. Prior to aneurysm treatment, with the patient already under general anesthesia, the blood supply to an arm will be restricted for 3x 5minutes by inflating a standard blood pressure cuff. The study hypothesis is that this "remote ischemic preconditioning" maneuver is able to prevent a stroke during the following treatment of the aneurysm.

DETAILED DESCRIPTION:
Prospective, randomized, double-blind, explorative single center clinical trial in patients subjected to the treatment of an un-ruptured intracranial aneurysm, either by surgical clipping or endovascular coiling. Goal of the study is to determine whether remote ischemic preconditioning (RIPC) prior to aneurysm treatment alters various biomarkers associated with ischemic central neuronal tissue damage. The trial takes place at Innsbruck University Hospital of Innsbruck Medical University, Innsbruck, Austria.

Patients fulfilling inclusion criteria are randomly allocated either to pre-interventional ischemic preconditioning (Group A = intervention group) or sham preconditioning (Group B = control group). RIPC is performed by inflating a blood pressure cuff around one upper extremity three times for five minutes with five minutes interval with the patient under general anesthesia prior to the start of the procedure.

Patients, all staff involved in diagnosis and treatment and all study members are blinded to the patients' group affiliation. The anesthesiologist and two staff members who perform preconditioning are not blinded.

Primary outcome is a difference of ± 2SD in the concentration-time curve of a panel of biochemical parameters indicative of cerebral ischemia (S100B, NSE, GFAP, MMP9, MBP, microparticles) in the first five days after the intervention. Secondary outcome parameters are changes in the post-interventional MRI and neuropsychological and clinical outcome at six and 12 months.

CONSORT and TIDieR guidelines will be followed. The trail will be registered in a public database. The trail protocol will be published in an open-access journal.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent of patient
* Age > 18 years
* Intracranial aneurysm, single or multiple, intervention as indicated by interdisciplinary vascular board (includes previously treated aneurysms)
* Normal baseline MRI

Exclusion Criteria:

* Clinical or radiological signs of subarachnoid hemorrhage
* Planned vessel sacrifice as the primary modality for aneurysm treatment
* Dissecting or mycotic aneurysm
* Previous history of stroke or TIA within the last six months
* Signs or symptoms of upper and lower extremity peripheral vascular illness
* Drugs and lifestyle factors that interfere with biomarker Determination
* Inability to complete neuropsychological testing for language reasons
* Patients unable to have an MRI scan for any reason
* Previous serious cerebral disease that would preclude completion of the protocol or preclude MRI analysis of small strokes
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Area-under-Curve for biomarkers in the first 5 days after aneurysm treatment(S100B, NSE, GFAP, NSE, MMP9, Microparticles) | on admission, after preconditioning but prior to intervention, at completion of intervention, at hours 3, 6, 12, 24, 48, 72, 96, 120 after completion of intervention
  Serum biomarkers reflect brain tissue ischemic damage with various specificity and sensitivity (see Whiteley 2008, Ahmad 2012) Advantages include (1) to be available early, (2) to be continuous variables (low study n), (3) they were able to demonstrate an effect of ischemic preconditioning in other clinical studies (see Koch 2010, Veighei 2012)

SECONDARY OUTCOMES:
Number (n) of new lesions in postinterventional MRI (DWI and FLAIR) | preinterventional/on day 1 or 2
  Outcome Parameter used in other clinical studies focussing on ischemia after neurointerventional procedures (e.g. ENACT study)
Clinical outcome ( National Institutes of Health Stroke Scale, NIHSS and modified Rankin Scale mRS) | at discharge, at 6 and 12 months
  Established outcome parameters for cerebrovascular studies. Dichotomized into favourable (NIHSS ≤1, mRS 0-1) and unfavourable
Volume (mm3) of new lesions in postinterventional MRI (DWI and FLAIR) | preinterventional, postinterventional on day 1 or 2
  As above for number of lesions

OTHER OUTCOMES:
Neuropsychological testing VLMTA (Verbaler Lern- und Merkfähigkeitstest), the WMS-R (Zahlenspanne vorwärts und rückwärts), trail making A and B tests, the Regensburger Wortflüssigkeitstest, the TAP Wechsel verbal, the TAP and the HADS-D) | preinterventional, at 6 and 12 months
  Standard tests used in patients with cerebrovascular disorders in our departments. Not applicable to non-german-speaking patients.
Brain volume changes (MRI, voxel -based morphometry) | Preinterventional/at the 12 months FU
  Longterm brain volume changes that correlate with NP deficits (Horstmann 2010, Moskowitz 2011, Vuylsteke 2011) will be analyzed using voxel-based morphometry techniques

CONTACTS AND LOCATIONS:
Overall Officials: Martin Ortler, M.D., MSc., Principal Investigator — Clinical Department of Neurosurgery, Innsbruck Medical University
Locations (1):
- Clinical Department of Neurosurgery, Innsbruck Medical University, Innsbruck, Austria